CLINICAL TRIAL: NCT04817553
Title: Impact of COVID-19 on the Clinical Outcomes and Management of IgG4 Related Disease Patients With Pancreatobiliary Involvement: a Multicenter Retrospective Study
Brief Title: Impact of COVID-19 on the Clinical Outcomes and Management of IgG4 Related Disease Patients
Acronym: IgG4-COVID
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond Shing Yan Tang, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: IgG4-COVID
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: IgG4 Related Disease; Covid19
Keywords: IgG4
MeSH Terms: conditions — Immunoglobulin G4-Related Disease; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IgG4 pancreatobiliary: IgG4 patients with pancreatobiliary involvement
  Interventions: Other: exposure to COVID19

INTERVENTIONS:
Other: exposure to COVID19 — Observational study of IgG4 patients with pancreatobiliary involvement who were diagnosed with COVID19

SUMMARY:
Since December 2019, coronavirus disease 2019 (COVID-19), caused by the severe respiratory syndrome coronavirus 2 (SARS-CoV-2), has affected more than 124 million people worldwide as of 23/3/2021. While studies on the outcomes of inflammatory bowel disease (IBD) (an important gastroenterological disease requiring immunosuppressive therapies for treatment) patients with COVID-19 have been published recently, little is known about the impact of COVID-19 on the clinical outcomes and management of IgG4 related disease patients with pancreatobiliary involvement. Because the number of IgG4 patients with pancreatobiliary involvement cared by individual centers and the prevalence of COVID-19 infection in different geographical regions vary, we propose to conduct a multicenter retrospective study to further evaluate the impact of COVID-19 on the clinical outcomes and management of IgG4 related disease patients with pancreatobiliary involvement.

DETAILED DESCRIPTION:
Since December 2019, coronavirus disease 2019 (COVID-19), caused by the severe respiratory syndrome coronavirus 2 (SARS-CoV-2), has affected more than 124 million people worldwide as of 23/3/2021. While many COVID-19 patients have been reported to have a milder clinical course, old age and comorbidities including cardiovascular disease, chronic lung conditions, obesity, and diabetes have been associated with a more severe disease course and higher mortality. Moreover, patients with chronic immune-mediated inflammatory diseases are at risk of viral infections either related to their underlying immune dysfunction or the immunosuppressive therapy that they receive for the chronic inflammatory conditions.

IgG4 related disease is an increasingly recognized immune-mediated condition that may resemble many malignant, infectious or inflammatory diseases. It is characterized by tumor-like lesions, with histopathological features of lymphoplasmacytic infiltrate rich in IgG4-positive plasma cells, obliterative phlebitis, storiform fibrosis, and, often but not always, elevated serum IgG4 concentrations.

While studies on the outcomes of inflammatory bowel disease (IBD) (an important gastroenterological disease requiring immunosuppressive therapies for treatment) patients with COVID-19 have been published recently, little is known about the impact of COVID-19 on the clinical outcomes and management of IgG4 related disease patients with pancreatobiliary involvement. Because the number of IgG4 patients with pancreatobiliary involvement cared by individual centers and the prevalence of COVID-19 infection in different geographical regions vary, we propose to conduct a multicenter retrospective study to further evaluate the impact of COVID-19 on the clinical outcomes and management of IgG4 related disease patients with pancreatobiliary involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or above
2. IgG4 related disease patients with pancreatobiliary involvement receiving care in the GI clinic of the participating centers
3. The diagnosis of IgG4 related disease was made either by:

   1. an elevated serum IgG4 serology level with typical features of pancreatobiliary involvement on imaging (eg, CT / MRI), and/or endoscopic ultrasound (EUS), and/or endoscopic retrograde cholangiopancreatography (ERCP), or
   2. an elevated serum IgG4 serology level with typical histopathologic features of the disease (eg, lymphoplasmacytic infiltration, obliterative phlebitis, and storiform fibrosis) on surgical pathology (eg, biopsy during surgery or surgical resection specimen) or endoscopic biopsies (eg, EUS guided fine needle biopsy).

Exclusion Criteria:

1) Patients who have an alternative diagnosis (i.e., non-IgG4 disease) despite an elevated serum IgG4 level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IgG4 patients with pancreatobiliary system involvement receiving care in the gastroenterology (GI) clinic in the participating centers fulfilling the inclusion criteria listed below and without exclusion criteria would be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Incidence of COVID-19 in IgG4 patients with pancreatobiliary involvement | Jan to Nov 2020
  Incidence of COVID-19 in IgG4 patients with pancreatobiliary involvement

SECONDARY OUTCOMES:
Incidence of severe COVID-19 in IgG4 patients with pancreatobiliary involvement | Jan to Nov 2020
  Incidence of severe COVID-19 in IgG4 patients with pancreatobiliary involvement (defined by the need of ICU admission, ventilator support, or death from COVID-19)
Medications for the underlying IgG4 disease used when patient was diagnosed to have COVID-19 | Jan to Nov 2020
  Medications such as steroid, steroid-sparing agents, biologics
Risk factors associated with COVID-19 infection in IgG4 patients with pancreatobiliary involvement | Jan to Nov 2020
  Risk factors include type of medication use, underlying medical conditions (such as diabetes, lung diseases, cardiovascular diseases, liver diseases)
Incidence of postponement or discontinuation of indicated medical treatment for the underlying IgG4 disease during COVID-19 outbreak | Jan to Nov 2020
  Incidence of postponement or discontinuation of indicated medical treatment for the underlying IgG4 disease during COVID-19 outbreak

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tang, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamisawa T, Zen Y, Pillai S, Stone JH. IgG4-related disease. Lancet. 2015 Apr 11;385(9976):1460-71. doi: 10.1016/S0140-6736(14)60720-0. Epub 2014 Dec 4. PMID 25481618